CLINICAL TRIAL: NCT03516175
Title: Pre-oxygenation With High-flow Nasal Cannula in Comparison to Standard in Adults During Rapid Sequence Induction Anesthesia- a Prospective Randomized Non-blinded International Multicenter Study
Brief Title: Pre-oxygenation With High-flow Nasal Cannula in Adults During Rapid Sequence Induction Anesthesia
Acronym: PRIOR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: St. George's Hospital, London (Other); University College London Hospitals (Other); Poole Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Senior Consultant, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIOR2
Record Dates: First submitted 2018-03-20; First posted 2018-05-04 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia; Hypoxia; Surgery; Acute
MeSH Terms: conditions — Hypoxia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight fitting mask (Active Comparator): Pre oxygenation with tight facemask with 100% oxygen
  Interventions: Device: Pre oxygenation using tight fitting facemask
- High flow nasal oxygen (Experimental): High flow nasal oxygen that is Transnasal Humidified Rapid Insufflation Ventilatory Exchange is used for pre oxygenation
  Interventions: Device: High flow transnasal oxygen

INTERVENTIONS:
Device: High flow transnasal oxygen — High flow nasal oxygen that is Transnasal Humidified Rapid Insufflation Ventilatory Exchange
  Other Names: Transnasal Humidified Rapid Insufflation Ventilatory Exchange
  Arms: High flow nasal oxygen
Device: Pre oxygenation using tight fitting facemask — 100% oxygen via a tight fitting facemask
  Arms: Tight fitting mask

SUMMARY:
It has been demonstrated that Transnasal Humidified Rapid Insufflation Ventilatory Exchange used during preoxygenation for emergency surgery is at least equally effective as preoxygenation compared to standard tight fitting mask. Data from a recent study indicates that Transnasal Humidified Rapid Insufflation Ventilatory Exchange might decrease the risk of clinically relevant desaturation below 93% of arterial oxygen saturation. The limitations with our previous study is that it was done only during office hours (Mon-Friday 8 am to 4 pm) and that the power to detect the occurrence of desaturation was too low.

Based on the above, the aim is now to conduct a clinical international multicenter study 24/7 with 450 patients and with a simplified protocol that allows the study to be done 24/7. This study is done with the aim of evaluation before implementing this novel technique of preoxygenation into clinical practice.

The general purpose of this project is to compare a the preoxygenation technique based on Transnasal Humidified Rapid Insufflation Ventilatory Exchange with traditional preoxygenation with a tight fitting mask during rapid sequence induction (RSI) intubation in patients undergoing emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, >18 years old
2. Emergency intubation where Rapid Sequence Induction is indicated
3. Capable of understanding the study information and signing the written consent.

Exclusion Criteria:

1. Body Mass Index >35
2. Pregnancy
3. Dependency on non-invasive ventilation to maintain oxygen saturation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
The number of patients that desaturates below 93% in SpO2 during pre oxygenation up to 1 minute after intubation | From start of anaesthesia until 1 minute after tracheal intubation, that is normally after 3-4 minutes after anaesthesia induction
  The number of patients that desaturates below 93% in SpO2 during pre oxygenation up to 1 minute after intubation

SECONDARY OUTCOMES:
Lowest SpO2 during preoxygenation using THRIVE compared to traditional pre-oxygenation from time to first anesthetic drug given up to 1 minute after intubation. | From start of anaesthesia until 1 minute after tracheal intubation, that is normally after 3-4 minutes after anaesthesia induction
  Lowest SpO2 during preoxygenation using THRIVE compared to traditional pre-oxygenation from time to first anesthetic drug given up to 1 minute after intubation.
Level of end-tidal carbon dioxide in the first breath after intubation with Transnasal Humidified Rapid Insufflation Ventilatory Exchange oxygenation compared with traditional pre-oxygenation? | At the first breath after tracheal intubation that is usually 2-4 minutes after induction of anaesthesia
  Level of end-tidal carbon dioxide in the first breath after intubation with Transnasal Humidified Rapid Insufflation Ventilatory Exchange oxygenation compared with traditional pre-oxygenation?
Level of end-tidal O2 in the first breath after intubation with Transnasal Humidified Rapid Insufflation Ventilatory Exchange oxygenation compared with traditional pre-oxygenation? | At the first breath after tracheal intubation that is usually 2-4 minutes after induction of anaesthesia
  Level of end-tidal O2 in the first breath after intubation with Transnasal Humidified Rapid Insufflation Ventilatory Exchange oxygenation compared with traditional pre-oxygenation?
Incidence of gastric regurgitation between the groups? | From start of anaesthesia until 2 minutes after tracheal intubation, that is normally after 4-5 minutes after anaesthesia induction
  Incidence of gastric regurgitation between the groups?
Difference in numbers of patients being ventilated between the two groups? | From start of anaesthesia until the patient is intubated, usually within 3-4 minutes
  Is there a difference in the number of patients that was ventilated before intubation between the two study groups?

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (6):
- Sweden (5):
  - Centralsjukhuset Karlstad, Karlstad
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
  - St Göran Hospital, Stockholm
  - Södersjukhuset, Stockholm
- University Hospital of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided